CLINICAL TRIAL: NCT02116998
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of GEN-004, a Pneumococcal Protein Subunit Vaccine, on Colonization Following Intranasal Challenge With S. Pneumoniae
Brief Title: Safety, Tolerability, and Efficacy Study of Prophylactic S. Pneumoniae Vaccine Following Challenge With S. Pneumoniae
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genocea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GEN-004-002; 2014-000944-13 (EudraCT Number)
Record Dates: First submitted 2014-04-11; First posted 2014-04-17 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Pneumococcal Infections; Pneumonia, Pneumococcal
Keywords: GEN-004; Aluminum hydroxide; Vaccine; Streptococcus pneumoniae; Pneumococcal Infections; Strep pneumoniae; Pneumonia
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia, Pneumococcal; Pneumonia | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GEN-004 with Aluminum Hydroxide (Experimental)
  Interventions: Biological: GEN-004 with Aluminum Hydroxide Adjuvant; Biological: Streptococcus pneumoniae inoculation
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo; Biological: Streptococcus pneumoniae inoculation

INTERVENTIONS:
Biological: GEN-004 with Aluminum Hydroxide Adjuvant — GEN-004: 100 µg of each antigen, with adjuvant, 350 µg aluminum hydroxide, administered as a 0.5 mL intramuscular (IM) injection.
  GEN-004 is a recombinant S. pneumoniae protein subunit vaccine consisting of 3 recombinant T cell antigens:
  * GB104: ABC transporter, substrate-binding protein
  * GB144: Maltose/maltodextrin binding protein, ABC transporter
  * GB152: Hypothetical protein
  GEN-004 is filled in 2 mL vials containing 0.5 mL (350 µg/mL of each antigen).
  Aluminum hydroxide adjuvant is filled in 2 mL vials containing 1 mL at a concentration of 5 mg/mL.
  Other Names: GEN-004
  Arms: GEN-004 with Aluminum Hydroxide
Biological: Placebo — Placebo: normal saline, 0.5 mL per dose, IM.
  Other Names: Saline; Normal saline
  Arms: Placebo
Biological: Streptococcus pneumoniae inoculation — Intranasal inoculation of S. Pneumoniae (80,000 CFU/100μl per nostril) serotype 6B.
  Other Names: S. Pneumoniae

SUMMARY:
This is a randomized, double-blind, placebo-controlled study. Eligible subjects will be randomized in a 1:1 ratio to receive GEN-004 with adjuvant or placebo. Each subject will receive up to 3 doses at 4 week intervals.

Following the third dose, subjects will be inoculated intranasally with S. pneumoniae serotype 6B. Nasal washes to identify S. pneumoniae colonization will be obtained pre-inoculation, and then 2, 7 and 14 days after inoculation.

Subjects will also be monitored for safety and tolerability throughout the dosing period, and then for 12 months after their last dose.

The purpose of this study is to evaluate the effectiveness of GEN-004 in reducing colonization rates and magnitude of colonization following the S. pneumoniae challenge.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females, ages 18 to 55 years inclusive.
* Willing and able to provide written informed consent.
* Fluent English speakers only (for safety reasons)
* Willing to perform and comply with all study procedures including attending clinic visits as scheduled.

Exclusion Criteria:

* Prior vaccination with pneumococcal vaccine.
* History of invasive pneumococcal disease (i.e., sepsis, meningitis or pneumonia with bacteremia).
* Close contact with at risk individuals (young children [under 5years], immunosuppressed adults, elderly, chronic ill health).
* Current smoker or significant smoking history (>10 pack years).
* Pregnant or breast-feeding woman.
* Women of child-bearing potential (WOCBP) who are deemed not to have sufficient, effective birth control in place for 1 month prior to vaccination and 1 month after the final vaccination.
* Allergy to penicillin or amoxicillin.
* Any screening laboratory value > Grade 1
* Positive serologic test for HIV-1 or hepatitis C infection; positive hepatitis B surface antigen (HBsAg).
* Asthma (on regular medication) or other respiratory disease.
* Immunocompromised individuals, including those receiving corticosteroids or other immunosuppressive agents.
* Presence or history of auto-immune disease (refer to Appendix 4) regardless of current treatment.
* No antibiotic treatment within 1 week of inoculation
* Previous involvement in EHPC study inoculated with pneumococcal bacteria
* In any other clinical trial unless in observational stage or follow-up
* Diabetes, type 1 or type 2.
* Other active, uncontrolled co-morbidities that, in the opinion of the Investigator would make the subject unsuitable for the study or unable to comply with the study requirements.

NOTE: Subjects who are taking a medication to control an underlying co-morbidity may be enrolled if there have been no changes to their medication within 60 days prior to first dose of Study Drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of GEN-004 with aluminum hydroxide in healthy adult subjects to reduce nasopharyngeal colonization following intranasal inoculation with S. pneumoniae serotype 6 as measured by proportion of colonized subjects | 56 weeks

SECONDARY OUTCOMES:
Safety and tolerability of GEN-004 with aluminum hydroxide | 56 weeks
Duration of S. pneumoniae colonization through 14 days after inoculation | 12 weeks
Immunogenicity of GEN-004 with aluminum hydroxide, as measured by TH17 (IL-17) and IgG responses to the vaccine antigens in sera and nasal fluid | 56 weeks
Impact of GEN-004 on the density of colonization as measured by S. pneumoniae colony forming units (CFUs) post-inoculation | 56 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Fitzgerald, MD, Principal Investigator — Royal Liverpool University Hospital
Locations (1):
- Royal Liverpool University Hospital, Liverpool School of Tropical Medicine, Liverpool, United Kingdom